CLINICAL TRIAL: NCT03005522
Title: The Effects of Dexamethasone on the Time to Pain Resolution in Dental Periapical Abscess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Noah Tolby, Principle Investigator, University of Arizona
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1611005004
Record Dates: First submitted 2016-12-24; First posted 2016-12-29 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Dental Research; Pharmaceutical Preparations, Dental
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): dosed with placebo
  Interventions: Drug: Placebo Oral Capsule
- intervention (Active Comparator): 10mg oral dexamethasone
  Interventions: Drug: oral dexamethasone

INTERVENTIONS:
Drug: oral dexamethasone — Patient will be dosed with either placebo or with the study drug, 10mg oral dexamethasone, to be administered by mouth one time in the ED
  Arms: intervention
Drug: Placebo Oral Capsule — dosed with placebo
  Arms: placebo

SUMMARY:
An individual's quality of life can be seriously affected by the severity of dental pain. The emergency department is a common place to find those seeking relief from their dental pain- often times seeking removal of the affected tooth, dental anesthetic injections or oral pain medications. There are a number of dental infections that cause this type of debilitating pain. One such dental infection is termed periapical abscess. This infection involves the tooth pulp. These infections can arise in three ways: introduction through a defect in the enamel and dentin; from a periodontal pocket or an adjacent tooth; or hematogenous seeding of the pulp from mechanical irritation. As this disease process continues there are a number of complications including chronic pain and, more seriously, the spread of infection into deep spaces which can be a life threatening condition.

The Emergency Department treatment of this infection includes pain control, antibiotics and dental referral for ultimate management of the infection.

The purpose of our study is to investigate whether the addition of oral steroids will alter the time until patient experiences improvement in their dental pain. Steroids are a commonly used anti-inflammatory that is used in the Emergency Departmentfor the purpose of pain relief from throat pain. As the pain from periapical infection is thought to be largely from the pressure we speculate that the anti-inflammatory effects of steroids may decrease the inflammation thus the pressure and may ultimately lead to a decrease in time until the patient experiences some relief from their pain.

ELIGIBILITY:
Inclusion Criteria:

Patients included if they had clinical diagnosis of pulpitis/dental apical abscess and physical exam revealed pain with percussion of the affected tooth/teeth plus or minus evidence of periapical abscess (gingival erythema, swelling, draining pus). Written informed consent was obtained from each patient prior to enrollment in the study.-

Exclusion Criteria:

1. Younger than 18 years old
2. Immunosuppression : HIV patient, transplant patient, chemotherapy
3. History of diabetes
4. Recent (<1 month) or chronic steroid use
5. Hospitalization required due to intractable vomiting/pain
6. Pregnancy, self report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Tolby, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Intervention
Started | 36 | 37
Completed | 25 | 27
Not Completed | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Intervention | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 52
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (10.8) | 33.9 (9.44) | 34.4 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 13 | 14 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants] — data not collected on race or ethnicity Population: data on race and ethnicity were not collected
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Decrease Time of Oral Pain
Description: The purpose of this study is to investigate whether the addition of oral steroids will alter the time until patient experiences improvement in their dental pain from an acute dental periapical abscess. The patients will be randomized to receive either dexamethasone or placebo. The patients will be contacted over a period 72 hours to assess their level of pain resolution.
  Pain was reported using a verbal numeric scale in which 10=maximum pain and 0=no pain
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 25 | 27
score on a scale
  At presentation | 9 [8 to 10] | 9 [8 to 10]
  At discharge | 5 [2 to 7] | 4 [2 to 7]
  At 12 hours | 5 [3 to 8] | 1 [0 to 5]
  At 24 hours | 3 [1 to 7] | 2 [0 to 5]
  At 48 hours | 3 [0 to 7] | 0 [0 to 2]
  At 72 hours | 1 [0 to 7] | 0 [0 to 2]

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Placebo | Intervention
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT03005522/Prot_SAP_000.pdf